CLINICAL TRIAL: NCT01175889
Title: Megadyne ACE Incision/Dissection Study
Acronym: ACE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Megadyne Medical Products Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ACE MS 1
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Abdominoplasty; Bilateral Breast Reduction; Bilateral Breast Lift; Bilateral Brachioplasty; Bilateral Lateral Thigh and Buttocks Lift

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- one side ACE blade (Experimental)
  Interventions: Device: E-Z Clean ACE Blade
- one side scalpel (Active Comparator)
  Interventions: Device: E-Z Clean ACE Blade

INTERVENTIONS:
Device: E-Z Clean ACE Blade — The prospective assessment of the E-Z Clean ACE electrosurgical electrodes using the ACE Blade in the ACE Mode for targeted procedures such as abdominoplasty, bilateral breast reduction, bilateral breast lifts, bilateral brachioplasty, bilateral lateral thigh and buttocks lifts, or any combination thereof.
  Other Names: ACE Blade

SUMMARY:
The Megadyne Ace™ Incision/ Dissection study is a post market, prospective assessment of the E-Z Clean ACE electrosurgical electrodes using the ACE Blade in the ACE Mode for targeted procedures such as abdominoplasty, bilateral breast reduction, bilateral breast lifts, bilateral brachioplasty, bilateral lateral thigh and buttocks lifts, or any combination thereof.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >18 years of age or < 60 years old
* Subject is undergoing abdominoplasty, bilateral breast reduction, bilateral breast lift, bilateral brachioplasty, bilateral lateral thigh and buttocks lift, or any combination thereof
* Subject is able to discontinue anticoagulant therapy (including Aspirin)
* Subject is willing and able to comply with study follow-up procedures
* Subject is willing to provide written informed consent for their participation in the study

Exclusion Criteria:

* Subject has a history of smoking in the last 6 months prior to surgery.
* Subject has a history of type I or type II Diabetes.
* Subject has an active infection of any kind at the time of enrollment
* Subject has a known coagulopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate Wound Healing/Scar Formation | 120 Days
  Primary Effectiveness Objective Evaluate wound healing/ scar formation between incisions made using a cold steel scalpel and incisions made using the ACE Blade per photographic evidence at 120 days by an independent observer

SECONDARY OUTCOMES:
Evaluate patient satisfaction relating to wound healing | 120 Days
  Secondary Effectiveness Objective Evaluate patient satisfaction relating to wound healing/ scar formation between incisions made using a cold steel scalpel and incisions made using the ACE Blade at 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Ryan D Lewis, M.D., Study Chair — Sponsor GmbH
Locations (3):
- United States (3):
  - Center for Plastic Surgery, Twin Falls, Idaho
  - Southwest Surgical Suites, LLC, Fort Wayne, Indiana
  - Plastic and Reconstructive Surgery University Health Sciences, Winston-Salem, North Carolina